CLINICAL TRIAL: NCT01394692
Title: Resection Control of Primary Brain Tumours Using a Low-Field Intraoperative MRI
Brief Title: Comparative Study of Intraoperative MRI-guided vs. Conventional Glioma Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Christian Senft, Neurosurgeon, Goethe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JWG-EK 239/07
Record Dates: First submitted 2011-07-13; First posted 2011-07-14 (Estimated); Results first posted 2012-11-28 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-10

CONDITIONS: Glioma
Keywords: intraoperative MRI; glioma surgery; extent of resection
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- intraoperative MRI (Active Comparator): tumor resection with intraoperative MRI-guidance
  Interventions: Procedure: intraoperative MRI-guided tumor resection
- conventional group (Active Comparator): standard microsurgical tumor resection
  Interventions: Procedure: standard microsurgery

INTERVENTIONS:
Procedure: intraoperative MRI-guided tumor resection — tumor resection with the use of an intraoperative MRI
  Other Names: PoleStar-N20 intraoperative MRI
  Arms: intraoperative MRI
Procedure: standard microsurgery — microsurgical tumor resection
  Arms: conventional group

SUMMARY:
Excision to the maximum possible extent marks the first step of glioma surgery. Depending on tumour histology, adjuvant treatment consists of radio- and/or chemotherapy. Multi-centre studies have shown that the presence of residual tumour according to MRI-criteria is a prognostic factor in this incurable condition.

In order to improve the extent of resection, several methods, in particular intraoperative imaging techniques, have become available to demonstrate already during surgery whether the goal of surgery has been achieved. The intraoperative MRI devices currently available differ in their magnetic field strengths and image resolution, but also in their amount of interference with the surgical workflow.

Prospective, high-class evidence data to promote the use of intraoperative MRI in glioma surgery are lacking. To assess whether the rate of radiologically complete tumour resections can be improved by using intraoperative MRI-guidance, we designed this prospective, randomized trial. We hypothesized that the extent of resection that can be achieved using an intraoperative MRI is greater than that of conventional microsurgical tumor resection.

ELIGIBILITY:
Inclusion Criteria:

* known or suspected contrast-enhancing glioma (primary and recurrent)
* location of the tumor permits intended gross-total resection

Exclusion Criteria:

* tumor location prohibits or questions gross-total resection
* contraindications to undergo MRI examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-10; Primary Completion 2010-07 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Senft, M.D., Principal Investigator — Goethe University; Volker Seifert, M.D., Study Director — Goethe University
Locations (1):
- Department of Neurosurgery, Goethe-University, Frankfurt, Germany

REFERENCES:
- [Result] Senft C, Bink A, Franz K, Vatter H, Gasser T, Seifert V. Intraoperative MRI guidance and extent of resection in glioma surgery: a randomised, controlled trial. Lancet Oncol. 2011 Oct;12(11):997-1003. doi: 10.1016/S1470-2045(11)70196-6. Epub 2011 Aug 23. PMID 21868284

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intraoperative MRI | Conventional Group
Started | 29 | 29
Completed | 29 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intraoperative MRI | Conventional Group | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 19 | 39
  >=65 years | 9 | 10 | 19
Age Continuous [Mean (Standard Deviation); unit: years] | 57 (13) | 58 (13) | 58 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 19 | 16 | 35
Region of Enrollment [Number; unit: participants]
  Germany | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Extent of Resection
Description: Number of patients with contrast-enhancing glioma in whom a complete excision of the tumor according to postoperative high-field MRI within 72 hours is achieved
Time Frame: 72 hours
Population: Patients in whom histological examination of tumor specimens did not result in diagnosis of a glioma were excluded for final analysis.
Measure: Number; unit: participants
Arm/Group | Intraoperative MRI | Conventional Group
Number analyzed (Participants) | 24 | 25
participants | 24 | 25

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (radiological and/or clinical progression) at 6 months following surgery
Time Frame: 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Volumetric Assessment
Description: Volumetric assessment of the extent of resection on early (within 72h) postoperative MRI
Time Frame: 72 hours
Reporting Status: Not Posted

4. Secondary Outcome: Neurological Deficit
Description: Assessment of new postoperative deficits following tumor surgery
Time Frame: 7 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Intraoperative MRI | Conventional Group
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 0/24 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes